CLINICAL TRIAL: NCT02850419
Title: Heat-Activated Target Therapy (Radiotherapy + Hyperthermia + Lyso-Thermosensitive Liposomal Doxorubicin) of Local-Regional Relapse in Breast Cancer Patients
Brief Title: Heat-Activated Target Therapy of Local-Regional Relapse in Breast Cancer Patients
Acronym: EURO-DIGNITY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-15-201
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ThermoDox (40mg/m2)+hyperthermia+RT (Experimental): Treatment will consist of up to six cycles of LTLD combined with hyperthermia every 21 days with the first day of each cycle being Day 1. ThermoDox will be administered at a dose of 40 mg/m2. Thermal dose is a one-hour treatment at a temperature between 40 and 43°C at the target site. At Cycle 1, radiotherapy will begin and will be combined with hyperthermia. A total of 40 Gy in 20 fractions of 2 Gy per fraction will be administered. Up to 66 Gy of radiation therapy can be administered however institutional guidelines should be followed.
  Interventions: Drug: ThermoDox (Thermally Sensitive Liposomal Doxorubicin); Radiation: Radiation Therapy; Device: Superficial Hyperthermia

INTERVENTIONS:
Drug: ThermoDox (Thermally Sensitive Liposomal Doxorubicin) — A dose of 40 mg/m2 will be administered at each cycle for a total of 6 cycles. ThermoDox will be administered in conjunction with hyperthermia.
Radiation: Radiation Therapy — A total of 40 Gy in 20 fractions of 2 Gy per fraction will be administered. Up to 66 Gy of radiation therapy can be administered however institutional guidelines should be followed.
Device: Superficial Hyperthermia — Thermal dose is an one-hour treatment at a temperature between 40 and 43 degrees Celsius at the target site.

SUMMARY:
The 105-15-201 study is designed to assess the effectiveness and tolerability of the combination of heat-activated target therapy (radiotherapy + hyperthermia + lyso-thermosensitive liposomal doxorubicin) of loco-regional relapse in breast cancer patients.

DETAILED DESCRIPTION:
Locoregional recurrence of breast cancer (LRR) after mastectomy is a clinically challenging problem. Between 5% and 35% of women with operable breast cancer will experience an isolated LRR following their primary treatment, usually within 5 years of initial mastectomy. LRR or LR typically causes pain, lymphedema, and/or loss of freedom of movement. Therapeutic options usually involve resection, radiation or, at some specialized centers, combined radiation and hyperthermia. However, local control remains suboptimal in previously irradiated chest wall patients with the combination of radiation and hyperthermia providing local control rates of about 65%.

Lyso-thermosensitive liposomal doxorubicin (LTLD) is a temperature sensitive liposome which is systemically administered and is engineered to selectively release its doxorubicin contents when exposed to temperatures ≥ 39.5°C.

Local mild hyperthermia (40 to 44°C) is cytotoxic and is known to have an immunomodulatory effect along with a radiation and chemosensitizing effect in the heated tissue. Furthermore, mild hyperthermia enhances leakiness of tumor tissue, increases local perfusion and upregulates transvascular transport of doxorubicin.

Radiation therapy will be administered in this combination therapy.

This study evaluates the application of a tri-modal approach with LTLD to improve outcome: radiation, hyperthermia, and targeted release of a novel formulation of doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented recurrent adenocarcinoma of the breast with a recurrence on the chest wall or its overlying skin:

   * Ulcerative chest wall disease defined as non-healing wounds consistent with cancer.
   * Inflammatory breast carcinoma.
   * Breast carcinoma not resected for medical reasons.
2. Tumor thickness, must be clinically indicated for hyperthermia therapy, as measured by clinical exam or radiological imaging studies (CT or MRI). The target local tumor lesion(s) must be able to be covered within two hyperthermia fields of treatment.
3. LRR Disease progression despite other available standard treatment options based on what is clinically indicated according to the investigator's clinical and medical judgment, including: one or more radiation treatment(s) to the chest wall
4. Patients with stable distant bone metastasis; concomitant treatment with Zoledronic acid and Denosumab is allowed
5. Non-pregnant female at least 18 years of age. If subject is of child-bearing age, must have a negative serum pregnancy test at baseline and must agree to practice an acceptable form of birth control while on the study.
6. Provide written informed consent and willing to comply with the protocol requirements.

Exclusion Criteria:

1. No concomitant cytotoxic antineoplastic therapy is allowed. Prior chemotherapy should not be administered within 5 half-lives or 28 days whichever is shorter.
2. Prior confirmed allergic reaction (including moderate rash, dyspnea, wheezing, urticaria or other symptoms) attributed to the administration of either anthracyclines or other liposomally encapsulated drugs that required discontinuation of prior therapy.
3. Patients who have previously received hyperthermia in conjunction with either radiation therapy or chemotherapy.
4. Previous treatment with anthracyclines exceeding the following dosages: free doxorubicin (i.e. non- liposomal) and/or liposomal doxorubicin ≥300 mg/m2 epirubicin free > 540 mg / m2.
5. Previous (required active treatment within 5 years) or concomitant malignancy except basal cell cancer, in situ carcinoma of the cervix, or contralateral breast cancer. Subjects with a prior contralateral breast malignancy can be included if they did not receive any chemotherapy.
6. Baseline laboratories (to establish eligibility): · Granulocytes ......< 1,500/ microliter · Platelets .......... < 75,000/ microliter · Hemoglobin ... < 9 gm/dL Total Bilirubin ... > 2 mg/dL ALT and AST ...> 2.5X upper limit of normal Creatinine ......... > 1.5 X upper limit of normal.
7. ECOG/Zubrod Performance Status > 2.
8. MUGA/Echocardiogram Left Ventricular Ejection Fraction < 50%.
9. History of: acute coronary syndrome, cerebral vascular accident, abnormal cardiac stress testing within last 6 months, symptomatic coronary artery disease, uncontrolled hypertension or cardiomyopathy and cardiac valvular surgery or open heart surgery.
10. Conditions which may interfere with hyperthermia portion of the trial such as: functioning cardiac pacemaker; metal plates, rods or prosthesis of the chest wall, breast reconstruction with implants, severe numbness and/or tingling of the chest wall or breast, skin grafts and/or flaps on the breast/CW.
11. Serious active infection requiring long-term antibiotic treatment.
12. Has received any external radiation therapy within 60 days prior to study enrollment.
13. Patients with parenchymal and known brain metastases; if metastasis is operated or irradiated the patient can be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 12 months
Loco-regional breast tumor control in patient who underwent ThermoDox + hyperthermia + radiotherapy as measured by target lesion clinical response rate combining RECIST criteria with digital photography to gauge response. | Up to 18 months

SECONDARY OUTCOMES:
Duration of local control [CR (complete response), PR (partial response) and SD (stable disease) following treatment with ThermoDox + Hyperthermia + Radiotherapy up to 12 months among patients with LRR breast cancer. | Up to 18 months
Patient Reported Quality of Life using the FACT-B following treatment with ThermoDox + Hyperthermia + Radiotherapy among patients with LRR breast cancer. | Up to 18 months
Patient Reported Quality of Life using the Brief Pain Inventory (BPI) following treatment with ThermoDox + Hyperthermia + Radiotherapy among patients with LRR breast cancer. | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Gabriele, M.D., Principal Investigator — FONDAZIONE DEL PIEMONTE PER L'ONCOLOGIA - IRCCS CANDIOLO
Locations (3):
- Inst. of Radiation Oncology Hospital Na Bulovce, Prague, Czechia
- Rambam Health Care Campus, Haifa, Israel
- Fondazione Del Piemonte Per L'Oncologia - Irccs Candiolo, Candiolo, Italy